CLINICAL TRIAL: NCT01067573
Title: The Role of Leptin Levels in Multiple Sclerosis
Brief Title: The Role of Serum Leptin Levels in Multiple Sclerosis Disease Activity While on Interferon Beta 1a (Rebif) Treatment
Acronym: Leptin
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Other Study IDs: USF 6175-A675E9
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2010-02

CONDITIONS: Multiple Sclerosis
Keywords: MS; Serum Leptin Levels during relapse; Multiple sclerosis; relapse
MeSH Terms: conditions — Multiple Sclerosis; Recurrence

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To determine a correlation between serum leptin levels, nitric oxide preceding a relapse and change in leptin and nitric oxide levels during exacerbation in relapsing remitting multiple sclerosis patients.

DETAILED DESCRIPTION:
This is an observational pilot study in patients with definitive relapsing-remitting multiple sclerosis to determine whether there is a correlation in serum leptin levels and serum nitric oxide levels during a clinically observed increase in disease activity. Each subject will followed for 12 months while taking interferon beta-1a subcutaneous injections 3 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple sclerosis per update of McDonald criteria
* Initiating treatment with interferon beta 1a subcutaneous injection with minimal dosing of 22mcg.
* 18-60 years of age.
* Women who are not pregnant or breast feeding, and who do not intend to become pregnant.
* Stable dose of concomitant medications for 30 days prior to baseline. Efforts should be made to maintain steady doses of concomitant medications for the duration of the study.

Exclusion Criteria:

* Treatment on other interferon preparations, glatiramer acetate, in last 30 days or 6 months on Natalizumab, mitoxantrone, cyclosporine or other immunomodulators as determined by the PI.
* Treatment with any other investigational treatments within the past year or treatment with any investigational treatments for multiple sclerosis within the last year.
* Any progressive form of MS.
* Known Hypersensitivity to interferon beta 1a.
* Inability to administer subcutaneous injections
* Inability to undergo laboratory evaluation.
* Seropositivity for HIV (by medical history)
* Diabetes Mellitus Tyle I or II (by medical history)
* Hepatitis B or C (by medical history)
* Uncontrolled psychiatric disorder.
* Any unstable illness that the investigator's opinion precludes participation in this study.
* Inability to maintain compliance with study protocol.
* Implanted devices or metal which would contraindicate MRI.
* Clinically significant abnormalities in CBC or CMP
* MMSE <25

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: USF Medical Clinic Tampa, Flrida
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-12; Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Fasting leptin and nitric oxide testing | monthly, for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J Krolczyk, DO, RPH, Principal Investigator — University of South Florida
Locations (1):
- USF Health, Tampa, Florida, United States

REFERENCES:
- [Background] De Rosa V, Procaccini C, La Cava A, Chieffi P, Nicoletti GF, Fontana S, Zappacosta S, Matarese G. Leptin neutralization interferes with pathogenic T cell autoreactivity in autoimmune encephalomyelitis. J Clin Invest. 2006 Feb;116(2):447-55. doi: 10.1172/JCI26523. Epub 2006 Jan 12. PMID 16410832
- [Background] Musio S, Gallo B, Scabeni S, Lapilla M, Poliani PL, Matarese G, Ohtsu H, Galli SJ, Mantegazza R, Steinman L, Pedotti R. A key regulatory role for histamine in experimental autoimmune encephalomyelitis: disease exacerbation in histidine decarboxylase-deficient mice. J Immunol. 2006 Jan 1;176(1):17-26. doi: 10.4049/jimmunol.176.1.17. PMID 16365391